CLINICAL TRIAL: NCT02663635
Title: Simulated Clinical Use Testing on Safe'n'Sound 1mL Staked Passive Delivery System With add-on Extended Finger Flanges
Brief Title: Simulated Clinical Use Testing on Safe'N'Sound 1ML Stalked Passive Delivery System With Add-On Extended Finger Flanges
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nemera La Verpilliere (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1550599
Record Dates: First submitted 2016-01-07; First posted 2016-01-26 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Needle Stick
MeSH Terms: conditions — Needlestick Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other)
  Interventions: Device: Safe'N'Sound

INTERVENTIONS:
Device: Safe'N'Sound

SUMMARY:
A simulated clinical use testing the Save'N'Sound 1mL staked Passive Delivery System with add-on extended finger flanges

DETAILED DESCRIPTION:
This study aims to evaluate the safety of the use of the Safe'N'Sound 1mL staked passive delivery system cone version with add-on EFF in the prevention of needle stick injuries and to evaluate the user's satisfaction with regards to the handling characteristics of the product namely safety, design and the ease of use.

ELIGIBILITY:
Inclusion Criteria:

The Evaluator must be:

* Minimum of age 18
* Able to understand and provide signed consent for the study
* Willing to comply with the study protocol, including being willing to answer questions and complete questionnaires
* Have no concerns about the ability to perform the simulated injections
* With no financial interest in the sponsor (Nemera) or the CRO (NAMSA)

Exclusion Criteria:

* If in the opinion of CRO, including the observer/monitor, the potential evaluator is not a good candidate for the study, including the reasons such as mental health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The true failure rate of the Safe'n'Sound 1mL Staked Passive Delivery system with add-on extended finger flange | At time of testing, day 1

SECONDARY OUTCOMES:
Ease of Use | At time of testing, day 1
Evaluator assessment of device handling | At time of testing, day 1
Evaluator assessment of instructions | At time of testing, day 1
Evaluator assessment of improvement of device over predecessor device | At time of testing, day 1

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pratt, Principal Investigator — NAMSA
Locations (1):
- NAMSA, Minneapolis, Minnesota, United States